CLINICAL TRIAL: NCT06776575
Title: Musculoskeletal Ultrasound and Electrophysiological Evaluation of the Hand in Patients With Systemic Sclerosis: Relation to Hand Dysfunction and Quality of Life
Brief Title: Ultrasound and Electrophysiology Study of Hand in Systemic Sclerosis Patients and Contributors of Hand Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Hossam Abdelrahman, Assistant Lecturer, Assiut University
Other Study IDs: hand ultrasound SSc patients
Record Dates: First submitted 2024-10-29; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Scleroderma; Hand Functionality; Quality of Life (QOL)
Keywords: hand dysfunction; musculoskeletal ultrasound; electrophysiology; quality of life; scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this research is to assess quality of life and hand function in systemic sclerosis patients via specific questionnaires, and to determine the main contributors to hand dysfunction via a thorough hand ultrasound study and electrophysiology study.

DETAILED DESCRIPTION:
Systemic Sclerosis (SSc) is a rare multiorgan autoimmune disease characterized by vasculopathy and fibrosis. Its prevalence rates vary greatly by geographic area from 9.3 to 660 per million.

The disease is primarily observed in individuals aged 35 to 55 years, with females being four to six times more affected than males. Hand involvement is an early manifestation of systemic SSc. It's recognized as a major driver of disability and diminished quality of life .

Managing hand pain can be particularly challenging due to the coexistence of non-inflammatory arthralgia, inflammatory arthritis, acro-osteolysis, tenosynovitis, joint contractures, tendon friction rubs, nerve entrapment, Raynaud's phenomenon, digital ulcers, sclerodactyly, calcinosis and chronic pain. Due to the multifactorial etiology of hand functional disability in SSc, it is important to define the contribution of each factor or structure to this issue. This understanding is essential for developing a rehabilitation and medical treatment oriented approach to disease management. While physical examination and radiographs are the first line methods for evaluating hand pain, they are limited in scope and miss many underlying etiologies of hand impairment.

Musculoskeletal ultrasound (MSUS) is rapidly becoming a mainstay diagnostic tool in the assessment of rheumatic diseases due to its low cost, portability, and safety as a non-ionizing imaging modality. The Outcome Measures in Rheumatology (OMERACT) Ultrasound working group has provided definitions for pathologic lesions seen in rheumatic disorders, which offers a valuable framework for the assessment of hand impairment in SSc.

ELIGIBILITY:
Inclusion Criteria:

Adult SSc Patients ( >18 yrs ) who are fulfilling the The EULAR/ACR 2013 classification criteria

Exclusion Criteria:

1. Individuals with other autoimmune diseases (systemic lupus, sjogren syndrome, rheumatoid arthritis dermatomyositis, mixed connective tissue disease).
2. Usage of drugs that can cause peripheral neuropathy and chronic alcohol abuse history.
3. Presence of diabetes mellitus, thyroid dysfunction and renal failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the Rheumatology, Rehabilitation and Physical medicine department, Assuit University hospitals. Informed consent will be obtained from all patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life in systemic sclerosis patients | 2 years
  Investigators will assess quality of life in systemic sclerosis patients using scleroderma health assessment questionnaire in order to help them improve their quality of life.
Hand function in systemic sclerosis patients . | 2 years
  Hand function in systemic sclerosis patients will be assessed using modified hand mobility score.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Duruoz MT, Poiraudeau S, Fermanian J, Menkes CJ, Amor B, Dougados M, Revel M. Development and validation of a rheumatoid hand functional disability scale that assesses functional handicap. J Rheumatol. 1996 Jul;23(7):1167-72. PMID 8823687
- [Result] Steen VD, Medsger TA Jr. The value of the Health Assessment Questionnaire and special patient-generated scales to demonstrate change in systemic sclerosis patients over time. Arthritis Rheum. 1997 Nov;40(11):1984-91. doi: 10.1002/art.1780401110. PMID 9365087
- [Result] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Result] Li L, Cui Y, Chen S, Zhao Q, Fu T, Ji J, Li L, Gu Z. The impact of systemic sclerosis on health-related quality of life assessed by SF-36: A systematic review and meta-analysis. Int J Rheum Dis. 2018 Nov;21(11):1884-1893. doi: 10.1111/1756-185X.13438. Epub 2018 Nov 14. PMID 30428506
- [Result] Tore NG, Sari F, Sarac DC, Baglan Yentur S, Satis H, Avanoglu Guler A, Haznedaroglu S, Oskay D. Inter-rater reliability of modified hand mobility in scleroderma test. Int J Rheum Dis. 2020 Feb;23(2):203-206. doi: 10.1111/1756-185X.13750. Epub 2019 Nov 19. PMID 31746119
- [Result] Sandqvist G, Nilsson JA, Wuttge DM, Hesselstrand R. Development of a modified hand mobility in scleroderma (HAMIS) test and its potential as an outcome measure in systemic sclerosis. J Rheumatol. 2014 Nov;41(11):2186-92. doi: 10.3899/jrheum.140286. Epub 2014 Oct 1. PMID 25274889
- [Result] Torok KS, Baker NA, Lucas M, Domsic RT, Boudreau R, Medsger TA Jr. Reliability and validity of the delta finger-to-palm (FTP), a new measure of finger range of motion in systemic sclerosis. Clin Exp Rheumatol. 2010 Mar-Apr;28(2 Suppl 58):S28-36. Epub 2010 Jun 10. PMID 20576211
- [Result] Aids to the Investigation of Peripheral Nerve Injuries. Revised second edition., Her Majesty's Stationery Office, 1943
- [Result] Merkel PA, Herlyn K, Martin RW, Anderson JJ, Mayes MD, Bell P, Korn JH, Simms RW, Csuka ME, Medsger TA Jr, Rothfield NF, Ellman MH, Collier DH, Weinstein A, Furst DE, Jimenez SA, White B, Seibold JR, Wigley FM; Scleroderma Clinical Trials Consortium. Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon. Arthritis Rheum. 2002 Sep;46(9):2410-20. doi: 10.1002/art.10486. PMID 12355489
- [Result] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Result] Bruyn GA, Iagnocco A, Naredo E, Balint PV, Gutierrez M, Hammer HB, Collado P, Filippou G, Schmidt WA, Jousse-Joulin S, Mandl P, Conaghan PG, Wakefield RJ, Keen HI, Terslev L, D'Agostino MA; OMERACT Ultrasound Working Group. OMERACT Definitions for Ultrasonographic Pathologies and Elementary Lesions of Rheumatic Disorders 15 Years On. J Rheumatol. 2019 Oct;46(10):1388-1393. doi: 10.3899/jrheum.181095. Epub 2019 Feb 1. PMID 30709946
- [Result] Silva A. M., Roque L. C, Gonçalves R. S, et al. Evaluation of quality of life, functionality and disability in patients with systemic sclerosis in a university hospital. ABCS Health Sci. 2020, 45, e020025.
- [Result] De Lorenzis E, Kakkar V, Di Donato S, Wilson M, Barnes T, Denton C, Derrett-Smith E, Douglas K, Helliwell P, Herrick AL, Saleem B, Nisar M, Morley C, Green L, Alcacer-Pitarch B, Del Galdo F. Clinical trajectories of hand function impairment in systemic sclerosis: an unmet clinical need across disease subsets. RMD Open. 2024 Jan 12;10(1):e003216. doi: 10.1136/rmdopen-2023-003216. PMID 38216288
- [Result] Caroline S. Morad, Reem A. Habeeb, Youssy S. et al. Hand and wrist musculoskeletal changes in systemic sclerosis patients, The Egyptian Rheumatologist, Volume 46, Issue 4, 2024
- [Result] Cevik R, Em S, Nas K, Toprak M, Cengiz G, Calis M, Sezer I, Unal Enginar A, Bora Karsli P, Sag S, Sargin B, Alkan Melikoglu M, Aydin Y, Duruoz MT, Gezer HH, Ecesoy H. Association of pain and clinical factors on disability and quality of life in systemic sclerosis: A cross-sectional study from Turkish League Against Rheumatism Network. Arch Rheumatol. 2022 Nov 11;38(1):9-21. doi: 10.46497/ArchRheumatol.2023.9243. eCollection 2023 Mar. PMID 37235112
- [Result] Balbach ML, Corty R, Hill B, Frech T, Aslam F, Chew EY. Development of a Musculoskeletal Ultrasound Protocol to Evaluate Hand Pain in Systemic Sclerosis Patients. Diagnostics (Basel). 2024 Mar 22;14(7):669. doi: 10.3390/diagnostics14070669. PMID 38611582